CLINICAL TRIAL: NCT00860353
Title: A Double Blind, Randomised, Placebo-controlled, Phase I Trial to Assess the Safety, Tolerability and Pharmacokinetics of Single, Ascending, Oral Doses of AZD2551 in Healthy Male Subjects
Brief Title: Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single Doses ofAZD2551
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to portfolio and logistical issues, this study will not be re-started at the present time. The study is not being terminated for safety reasons.
Sponsor: AstraZeneca (Industry)
Responsible Party: Harsukh Parmar MD, ChB, Global Head of Early Development, Respiratory and Inflammation Area, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D1570C00001
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: Healthy Volunteer; Single Ascending Dose; Safety; Tolerability; AZD2551; Healthy Volunteer Study

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD2551
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2551 — Single dose of oral solution.
  Arms: 1
Drug: Placebo — Single dose of oral solution
  Arms: 2

SUMMARY:
The purpose of this study is to determine how well tolerated and safe AZD2551 is at different dose levels in healthy, non-smoking males. It will also investigate how quickly AZD2551 is absorbed into and cleared by the body

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated informed consent prior to any study specific procedures
* Be willing to use barrier methods of contraception unless their partners are post-menopausal, surgically sterile or using accepted contraceptive methods
* Have a body mass index between 18 and 30 kg/m2 inclusive and weight at least 50kg and no more than 100kg

Exclusion Criteria:

* Use of any prescribed or non-prescribed medication during the two weeks prior to the administration of study drug
* History or presence of conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs
* Any impairment of kidney function or laboratory results for markers of kidney function that are outside the reference range and considered clinically significant
* Underlying musculoskeletal symptoms of unknown origin, subjects with shoulder girdle musculoskeletal symptoms or Dupuytrens syndrome

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-02; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AZD2551 by assessment of vital signs, ECG, laboratory variables and adverse events | Baseline assessments at Visit 1 (enrolment). Assessments pre-dose and at defined timepoints post-dose at Visit 2. Follow up assessment at Visit 3
Pharmacokinetic profile: concentration of AZD2551 in blood | Samples taken at Visit 2. Up to 15 samples to be taken at defined timepoints post-dose, plus one sample pre-dose

SECONDARY OUTCOMES:
Pharmacokinetic profile: concentration of AZD2551 in urine | Samples collected at Visit 2 from pre-dose up to 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: William Fahy, MA, MBBS (Hons), Principal Investigator — AstraZeneca Clinical Pharmacology Unit, E Floor, Queens Medical Centre, Nottingham NG7 2UH
Locations (1):
- Research Site, Nottingham, United Kingdom